CLINICAL TRIAL: NCT03981991
Title: Assessment of the Quality of Life for Patients Suffering From Isolated Endometriosic Lesion of Utero-sacral Ligaments Diagnosed by MRI, Before and After Surgical Treatment by Using French Version of Endometriosis Health Profile 30 (EHP30)
Brief Title: Endometriosis and Quality of Life Assessed by EHP 30
Acronym: ENDOLUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.130; 2019-A01143-54 (Other: ID RCB)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Endometriosis
Keywords: EHP 30; Endometriosis; Quality of Life; Uterosacral Ligament
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the quality of life for patients suffering from isolated endometriosic lesion of utero-sacral ligaments diagnosed by MRI, before and after surgical treatment by using French version of Endometriosis Health Profile 30 (EHP 30).

This is prospective, non-controlled, non-randomized, monocentric, observational feasibility study.

DETAILED DESCRIPTION:
Endometriosis is a gynecological pathology affecting women during periods of genital activity, which prevalence is underestimated and varies from 10 to 30%. It is characterized by dysmenorrhea, dyspareunia, chronic pelvic pain or infertility. These various manifestations lead to an alteration of the quality of life.

Among women consulting for chronic pelvic pain or suspicion of endometriosis, it is recommended to evaluate pain, as well as suggestive symptoms and localizers using validated quality of life questionnaires such as Endometriosis Health Profile 30 (EHP 30).

In case of chronic pelvic pain and suspicion of a deep lesion, the assessment of disease is based on the interrogation (deep and positional dyspareunia, urinary or digestive catamenial functional signs), pelvic clinical examination by a referral physician, an endovaginal ultrasound by a referral sonographer and pelvic MRI also by a referral radiologist.

However, interpretation is not always easy with a high rate of false negatives. In case of absence of pathognomonic iconographic signs and, if there is an impact on patients' quality of life, a diagnostic laparoscopy can be proposed. This procedure can help to affirm or invalidate endometriotic lesions not visible in imaging, allowing either an excision or lesion destruction.

Although the beneficial role of surgical management in spontaneous fertility has been demonstrated, the clinical benefit of reducing pain and improving the quality of life in isolated uterine sacral ligament lesions has not been demonstrated by clinical studies with a good level of evidence.

Through this study, we would like to evaluate the functional benefit on the quality of life in the short and medium term of laparoscopic surgical management in case of suspicion of isolated uterosacral ligament endometriosis documented by standardized pelvic MRI.

All MRI exams will be analyzed blindly by an expert radiologist.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged from 18 to 50 years
2. Patient with medical sign proving endometriotic lesion: dysmenorrhea, deep dyspareunia or chronic pelvic pain
3. Patient with standardized pelvic MRI realized at CHUGA
4. Patient with an indication for laparoscopic surgical treatment
5. Patient available to complete the questionnaire based on EHP 30
6. Patient available for a follow-up of 6 months
7. Patient able to understand and read French language
8. Patient affiliated to a social security system or beneficiary of the same.
9. Patient who agreed to participate to the research

Exclusion Criteria:

1. Patient with functional urinary or digestive signs related to endometriotic lesion
2. Patient with another deep lesion proved by MRI: endometrioma, rectovaginal septum, recto-sigmoid, urinary bladder, ureters, recto-uterine pouch.
3. Virgin patient
4. Patient with a contraindication to MRI
5. History of extensive pelvic surgery related to endometriosis
6. Pregnancy
7. Patient who did not receive laparoscopic treatment of uterosacral ligaments
8. Patient already involved in another clinical research study
9. Patient in a period of exclusion from another clinical research study
10. Referred to the Articles L1121-5, L1121-6, and L1121-8 of the Public Health Code (corresponds to protected persons: pregnant woman, parturient, breastfeeding mother, person deprived of liberty by judicial or administrative decision, legally protected subject).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women during periods of genital activity with medical sign proving endometriotic lesion of utero-sacral ligaments: dysmenorrhea, deep dyspareunia or chronic pelvic pain referred to Obstetrics and Gynecological Department of University Hospital of Grenoble
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Assess the quality of life of patients before and 3 months after laparoscopic treatment of isolated endometriosic lesions of uterosacral ligaments by French version of the EHP 30 questionnaire. | 3 months
  Overall score and scores by subdomains of EHP 30 questionnaire preoperatively and at 3 months postoperatively.

SECONDARY OUTCOMES:
Evolution of EHP 30 score (and its subdomains) preoperatively, and at 1, 3 and 6 months postoperatively. | 1 , 3 and 6 months
  Overall score, and scores by subdomains, of EHP 30 questionnaire at 1, 3 and 6 months postoperatively.
Assess diagnostic performances of MRI for diagnosis of lesions of uterosacral ligaments by correlating MRI's results with those of laparoscopy. | 1 month
  Uterosacral ligaments (yes / no) on MRI vs. laparoscopy.
Correlate, a posteriori, MRI results with findings of laparoscopy and EHP 30 score evolution | 3 months
  Uterosacral ligaments (yes / no) on MRI vs overall score of EHP 30 questionnaire preoperatively and at 3 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry MICHY, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France